CLINICAL TRIAL: NCT06001164
Title: Double-bundle Versus Single-Bundle Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Study With 15-Year Results
Brief Title: Double-bundle Versus Single-Bundle Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Arttu Seppanen, Principal Investigator, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R20001
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-bundle (Active Comparator)
  Interventions: Procedure: ACL reconstruction: Double bundle
- Single-bundle (Active Comparator)
  Interventions: Procedure: ACL reconstruction: Single bundle

INTERVENTIONS:
Procedure: ACL reconstruction: Double bundle — DB: Two tunnels were created on the femoral side through an anteromedial portal. These tunnels were created manually. On the tibial side, the tunnels were created using a guide to ensure they matched the anatomic insertion site of the ACL at the tibia. The hamstring grafts for the procedure were then harvested from the same leg and doubled. The femoral side was fixed from the inside out, whereas the tibial side was fixed from the outside in. bioresorbable screws were used.
  Arms: Double-bundle
Procedure: ACL reconstruction: Single bundle — SB: The femoral tunnel was created using an anteromedial portal. A freehand technique was used. For the tibial tunnel, a tibial guide was used to ensure it was positioned at the midpoint of the tibial ACL attachment site. The tendons of the semitendinosus and gracilis muscles were then harvested, doubled over, and inserted through the tibial tunnel, extending into the femur, and fixed with metallic or bioabsorbable interference screws.
  Arms: Single-bundle

SUMMARY:
The purpose of this study is to compare double-bundle and single-bundle techniques for ACL reconstruction in a long-term 15-year follow-up. Our hypothesis is that the DB technique is better than the SB technique.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients had to meet certain criteria, including primary ACL reconstruction, closed growth plates, and no ligamentous injuries to the contralateral knee.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
osteoarthritis (OA) | 15 years
  which group has more osteoarthritis? Kellgren Lawrence classification. Scale 0-4 (0=no OA)
Pivot shift | 15 years
  which group has more positive pivot shift tests? Always compared to a "healthy" knee.
KT-1000 arthrometer difference | 15 years
  Anteroposterior translation. Always compared to a "healthy" knee. mm.
Lysholm score | 15 years
  subjective evaluation form. Scale 0-100 (100=best)
IKDC subjective evaluation. Scale 0-100 (100=best) | 15 years
  subjective evaluation form
IKDC objective score. Scale 1-4 (1=best) | 15 years
  Overall evaluation of the knee
graft failures | 15 years
  which group has more graft failures? The number of graft failures was assessed by revision surgery.
Range on motion (ROM) of the knee | 15 years
  Which group has more lack of knee extension or lack of knee flexion? Injured knee is always compared to a contralateral "healthy" knee. Measurements were performed with a goniometer. ROM included lack of passive extension (normal < 3°, nearly normal 3-5°, abnormal 6-10°, and severely abnormal > 10°) and lack of passive flexion (normal 0-5°, nearly normal 6-15°, abnormal 16-25°, and severely abnormal > 25°).
One leg hop test | 15 years
  One leg hop test was performed to assess the functional capacity of the knee. The patient hopped a maximum length three times on each leg separately and the best result was recorded for both legs. The result of the operated leg was then compared with that of the non-operated leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics, Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No